CLINICAL TRIAL: NCT02551484
Title: Contribution of Near-InfraRed Spectroscopy (NIRS) to the Evaluation of Microcirculation Following Trans-tibial Amputation for Peripheral Artery Disease
Brief Title: Contribution of Near-InfraRed Spectroscopy (NIRS) to the Evaluation of Healing After Amputation of the Leg
Acronym: NIRS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The patient population presenting in the department has evolved and no longer allows for the recruitment of the necessary number of patients.
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CASILLAS Fd. Avenir 2012
Record Dates: First submitted 2015-08-20; First posted 2015-09-16 (Estimated); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: A Stabilized Definitive Prosthesis (Procedure 1); Definitive Prosthesis With a Contact Socket (Procedure 1); Patients in the Initial Phase (Temporary Prosthesis, Rehabilitation) Following Unilateral Post- Transtibial Amputation (Procedure 2)

ARMS (2):
- Procedure 1 (Experimental): Measures with 60 minutes interval during the consultation of equipment, functional testing, receuil pain.
  Interventions: Device: Measurements using NIRS; Device: TCPO2 measurements; Other: 2-minute walk test
- Procedure 2 (Experimental): Measuring J15, J30 J 45 and after the different settings functional amputation, pain and tissue oxygenation.
  Interventions: Device: Measurements using NIRS; Device: TCPO2 measurements

INTERVENTIONS:
Device: Measurements using NIRS
Device: TCPO2 measurements
Other: 2-minute walk test
  Arms: Procedure 1

SUMMARY:
50 patients will be included for each of the 2 procedures:

- For procedure 1: Patients will be selected during multidisciplinary consultations for amputees who are stabilized with their definitive prosthesis and have returned to their usual place of residence. The aim of this procedure is to show the validity and reproducibility of measurements of tissue oxygenation using NIRS (TcPO2 being the reference measurement), to determine the way in which NIRS measurements are more precise (i.e. in terms of validity and reproductibility) (values at rest with the patient lying perfectly flat or with the amputated limb raised 30°). These patients will require a single visit which will include measurements by NIRS and TCPO2, a walk test and the completion of 2 questionnaires (visual scale).

- For procedure 2: The patients will be included in the initial phase of postamputation rehabilitation, during the period of in-hospital rehabilitation. The main problems of healing and tolerance to the temporary prosthesis arise during this phase. The specific objectives will be: To show that measurement by NIRS predicts the quality of healing in trans-tibial amputees; to show that the zone of uncertainty concerning the predictive values for the viability of the stump is smaller with NIRS than with TcPO2 (better discrimination). NIRS and TCPO2 measurements as well as the evaluation of stump healing will be done 15, 30 and 45 days after the amputation.

ELIGIBILITY:
Inclusion Criteria:

All groups:

* Patients who have agreed to take part in the study
* Patients with National Health Insurance cover,
* Patients (men or women aged between 18 and 85 years, presenting unilateral transtibial amputation for PAD.
* Able to understand simple instructions

Procedure 1:

* Stabilized patients with their definitive prosthesis, with no modification of the prosthesis in the previous 3 months and at least 6 months after the amputation.
* Definitive prosthesis with a contact socket.
* Patients able to do a 2-minute walk test.

Procedure 2:

- Patients in the initial phase of post-amputation (temporary prosthesis, rehabilitation) following unilateral transtibial amputation.

Exclusion Criteria:

* Patients without national health insurance cover.
* Patients under guardianship.
* Patients with associated chronic motor deficiency, of a neurological origin (examples: sequelae of stroke, balance and coordination disorders), or osteo-articular disease (examples: knee or hip osteoarthritis), given their secondary functional impact, making it impossible for amputees to walk with a prosthesis.
* Severe medical disorder that significantly impairs functional abilities (severe heart failure, respiratory failure, non-stabilized metabolic disorders, such as progressive kidney failure) and diseases with an impact on short or medium-term survival (progressive neoplastic disease, non-stabilized systemic disease).
* Complications, other than microcirculatory, with the stump, able to affect the use of a contact socket: hematoma, formation of cysts, fluid build-up, calcifications of soft tissues, bone spur, infection (skin, abscess), neurinoma, deterioration of the knee joint of the amputated limb, angle of the tibial cut leading to specifically painful osteo-cutaneous impingement, venous thrombosis, abnormal shape of the stump making it unsuitable for a socket (flexum of the knee, "pear shaped" stumps or stumps with severe invaginations )…
* Local skin disorders in the measurement zone (summit of the antero-external area) of the stump compromising the quality of the signals picked up by the electrode (NIRS and TcPO2) : severe edema, hyperkeratosis, ulceration, inflammatory and infectious phenomena.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2013-01-15 (Actual); Primary Completion 2018-11-16 (Actual); Study Completion 2018-11-16 (Actual)

PRIMARY OUTCOMES:
For procedure 1: the intra-class correlation coefficient between two successive NIRS measurements. | Baseline
For procedure 1: the Cronbach alpha coefficient between the NIRS and TcPO2 measurements (the latter being the gold standard). | Baseline
For procedure 2: NIRS values at the first consultation and the time to complete healing. | Up to 60 days
Procedure 2: NIRS values measured at different sessions and the associated healing evaluation. | 45 days after the amputation

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de DIJON, Dijon, France

REFERENCES:
- [Result] Laroche D, Barnay JL, Tourlonias B, Orta C, Obert C, Casillas JM. Microcirculatory Assessment of Arterial Below-Knee Stumps: Near-Infrared Spectroscopy Versus Transcutaneous Oxygen Tension-A Preliminary Study in Prosthesis Users. Arch Phys Med Rehabil. 2017 Jun;98(6):1187-1194. doi: 10.1016/j.apmr.2016.12.001. Epub 2016 Dec 31. PMID 28049004